CLINICAL TRIAL: NCT01146808
Title: Prevention of de Novo Hepatitis B Infection With Adefovir Dipivoxil (ADV) and Hepatitis B Vaccination in HBsAg Seronegative Recipients of Liver Grafts From Hepatitis B Core Antibody Positive (HBcAb+) Donors
Brief Title: Adefovir Plus Vaccination in Transplant Patients Without Hepatitis B That Receive a Core Antibody Positive Liver
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB8413; IN-US-103-0158 (Other: Gilead)
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B; Liver Transplantation
Keywords: Vaccination; Immunocompromised Host; Antiviral Agents; Drug Resistance, Viral; Resource Allocation
MeSH Terms: conditions — Hepatitis B | interventions — adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADV plus hepatitis B vaccination (Experimental): Adefovir dipivoxil and hepatitis B vaccination: All subjects will receive adefovir 10mg po daily, or adjusted for renal function and an option for Hepatitis B vaccination, double dose.
  Interventions: Drug: Adefovir dipivoxil and hepatitis B vaccination

INTERVENTIONS:
Drug: Adefovir dipivoxil and hepatitis B vaccination — Adefovir 10mg po daily, or adjusted for renal function and option for Hepatitis B vaccination, double dose
  Other Names: Hepsera

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of adefovir (ADV) in preventing de novo Hepatitis B in patients who receive Hepatitis B core antibody (HBcAb) positive grafts but who are not Hepatitis B Surface antigen (HBsAg) positive prior to transplant (Hepatitis B naive patients). The second objective is to evaluate the efficacy of accelerated vaccination with Hepatitis B in inducing innate immunity, thereby obviating the need for life-long antiviral therapy.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, open-label study of Hepatitis B naive patients who received HBcAb + livers and adefovir prophylaxis post-transplant. At one year to 18 months following transplantation, all study patients will then be vaccinated with standard Hepatitis B vaccine at double dose on a monthly basis for three months, at which point they will be tested for Hepatitis B surface antibody (HBsAb). Any study patients that have developed a sufficient antibody response (HBsAb >500 IU) will be given the option to discontinue anti-viral treatment in a monitored setting.

ELIGIBILITY:
Inclusion Criteria:

* Recipients who do not have evidence of hepatitis B surface antigen, regardless of HBcAb and HBsAb status, who:

  1. received liver transplantation with hepatitis B core antibody positive (and HBsAg negative) grafts,
  2. received adefovir treatment post transplantation, and
  3. who have not reached the 18 month post transplantation time period.

Exclusion Criteria:

* Recipients with hepatitis B surface antigen positivity prior to liver transplant.
* Grafts from hepatitis B surface antigen positive patients.
* Previous intolerance to ADV therapy
* Recipients with pre-transplant creatinine > 1.6 mg/dL
* Patients younger than 21 years of age
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Brown, Jr, MD, MPH, Principal Investigator — Center for Liver Disease and Transplantation at Columbia University Medical Center
Locations (1):
- Center for Liver Disease and Transplantation at Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wachs ME, Amend WJ, Ascher NL, Bretan PN, Emond J, Lake JR, Melzer JS, Roberts JP, Tomlanovich SJ, Vincenti F, et al. The risk of transmission of hepatitis B from HBsAg(-), HBcAb(+), HBIgM(-) organ donors. Transplantation. 1995 Jan 27;59(2):230-4. PMID 7839446
- [Background] Saab S, Chang AJ, Comulada S, Geevarghese SK, Anselmo RD, Durazo F, Han S, Farmer DG, Yersiz H, Goldstein LI, Ghobrial RM, Busuttil RW. Outcomes of hepatitis C- and hepatitis B core antibody-positive grafts in orthotopic liver transplantation. Liver Transpl. 2003 Oct;9(10):1053-61. doi: 10.1053/jlts.2003.50208. PMID 14526400
- See also: Liver Transplantation information from the NIH — http://www.nlm.nih.gov/medlineplus/livertransplantation.html

RESULTS

PARTICIPANT FLOW:
Groups:
- ADV Plus Hepatitis B Vaccination Group: This group included recipients of Hepatitis B Core Antibody Positive livers who are negative for Hepatitis B infection.
Period: Overall Study
Arm/Group | ADV Plus Hepatitis B Vaccination Group
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ADV Plus Hepatitis B Vaccination Group
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Development of de Novo Hepatitis B Infection After Transplant With a Core Antibody Positive Liver
Description: Determined by positive hepatitis B serology (tests positive for HBsAg) and HBV DNA viral load (>40 IU/mL).
Time Frame: Standard of care visits post-transplant for 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ADV Plus Hepatitis B Vaccination Group
Number analyzed (Participants) | 16
Participants | 5

2. Secondary Outcome: Proportion of Patients With a Sustained Hepatitis B Surface Antibody Titer > 500 IU/mL Prior to and After Vaccination
Time Frame: 12-18 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | ADV Plus Hepatitis B Vaccination Group
Number analyzed (Participants) | 16
Participants | 2

3. Secondary Outcome: Proportion of Patients Who Develop de Novo Hepatitis B Infection Post ADV Withdrawal, Which Will be Assessed at 6 Months Post Withdrawal
Time Frame: Six months after hepatitis B vaccination (2 years post transplant)
Measure: Count of Participants; unit: Participants
Arm/Group | ADV Plus Hepatitis B Vaccination Group
Number analyzed (Participants) | 16
Participants | 3

ADVERSE EVENTS:
Arm/Group | ADV Plus Hepatitis B Vaccination Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No